CLINICAL TRIAL: NCT05999604
Title: Impact of Annual Versus Biannual Infusions of Ocrelizumab in Patients With Active MS,After 2 Years of Initial Treatment, on Freedom From Radiological Disease Activity at Two Years: a Multicenter Randomized Controlled Non-inferiority Trial
Acronym: WINDOCRE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBR_2022_13
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- annual ocrelizumab infusions (Experimental)
  Interventions: Drug: Ocrelizumab Injection [Ocrevus]
- semestrial ocrelizumab infusions (Other)
  Interventions: Drug: Ocrelizumab Injection [Ocrevus]

INTERVENTIONS:
Drug: Ocrelizumab Injection [Ocrevus] — Semestrial administration
  Arms: semestrial ocrelizumab infusions
Drug: Ocrelizumab Injection [Ocrevus] — Annual administration
  Arms: annual ocrelizumab infusions

SUMMARY:
Multiple sclerosis (MS) is a chronic autoimmune disease of the central nervous system and the leading cause of severe non-traumatic disability in young people, affecting 110,000 people in France. Ocrelizumab, a humanized anti-CD20 monoclonal antibody, has shown remarkable efficacy in Phase III trials on the inflammatory component of the disease, reducing the annualized relapse rate by 46% and the rate of new T2 lesions by 80% compared with interferon-β 1a.

The use of anti-CD20 agents, including ocrelizumab, is associated with an infectious risk that increases with duration of exposure, part of which is due to the development of hypo-gammaglobulinemia in relation to cumulative dose.

Several reports suggest a persistent effect of anti-CD20 drugs in MS, with no resumption of inflammatory activity after discontinuation:

* During the development of ocrelizumab, at the end of phase 2, after having received 3 or 4 semi-annual cycles of ocrelizumab, a safety period with a therapeutic window of 18 months was planned, before re-administration in the extension study. During this therapeutic window, the annualized relapse rate remained stable, and patients showed no radiological disease activity.
* Scandinavian observational studies of "off-label" use of anti-CD20 in MS provide real-life evidence of the absence of recovery of clinical and radiological activity after prolonged interruption of treatment.

After 2 years of treatment, and with disease activity under control, spacing administration intervals could reduce the risk of infection without reducing treatment efficacy. This would facilitate the decision to maintain highly active immunotherapy over the long term. In addition, this therapeutic de-escalation, by reducing the frequency of infusions and associated day hospitalizations, would help to reduce treatment management costs.

Our aim is to evaluate the non-inferiority of 12-monthly spacing of ocrelizumab infusions versus the conventional 6-monthly regimen, in a population of active MS patients over 18 years of age who have already received 4 or more semi-annual cycles of treatment for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 18 years of age or older
2. Presenting for a 4th semi-annual cycle of ocrelizumab (minimum)
3. Requires follow-up MRI as part of treatment.
4. Initial indication for ocrelizumab according to the marketing authorization (active MS, RR or SP form)
5. Absence of relapse for at least 18 months (a relapse being defined as the appearance of new symptoms or worsening of existing symptoms, lasting more than 24 hours and outside a period of fever or an infectious episode; notified as a validated relapse by the neurologist in the patient's file, treated or not with boluses of Solu-Medrol).
6. EDSS between 0 and 6 inclusive
7. Having received informed information about the study and having signed a consent to participate in the study
8. French language proficiency
9. Affiliated or beneficiary of a social insurance scheme

Exclusion Criteria:

1. Clinical forms of primary progressive MS
2. Patients already receiving systematically spaced doses of ocrelizumab ≥ 9 months apart
3. Contraindication to continued treatment with ocrelizumab (hypersensitivity reaction, ongoing active infection, development of malignancy since previous injection, development of severe immune deficiency)
4. Planned pregnancy within 3 years
5. Contraindication to MRI
6. Contraindication to injection of contrast media
7. Subject with severe or uncontrolled symptoms of renal, hepatic, hematological, gastrointestinal, pulmonary, psychiatric or cardiac disease, or any uncontrolled intercurrent pathology.
8. Patient under legal protection
9. Patients of childbearing age who do not wish to use effective contraception
10. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Absence of radiological disease activity at 2 years | Months24
  Percentage of patients with no new or enlarged T2 lesion >3mm on cerebrospinal MRI at 24 months compared with inclusion MRI.
  MRI readings at inclusion and M24 will be performed by an independent radiologist blinded to the treatment arm.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Hôpital Henri Mondor, Créteil
  - CH Gonesse, Gonesse
  - CHU de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - Hôpital Pierre Wertheimer (HCL), Lyon
  - CHU de Nice, Nice
  - Hôpital de la Pitié-Salpêtrière, Paris
  - Fondation Adolphe de Rothschild, Paris
  - CHI Poissy-Saint-Germain en Laye, Poissy
  - CHU de Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No